CLINICAL TRIAL: NCT06249438
Title: An Exploratory Clinical Study of Cluster of Differentiation Antigen 20(CD20)/Anti-B-cell Maturation Antigen(BCMA) Chimeric Antigen Receptor Autologous T Cell Product (C-CAR168) in the Treatment of Autoimmune Diseases Refractory to Standard Therapy
Brief Title: A Study of C-CAR168 in the Treatment of Autoimmune Diseases Refractory to Standard Therapy
Acronym: CAR-AID
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: AbelZeta Pharma Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1141-043(CAR-AID)
Record Dates: First submitted 2024-01-21; First posted 2024-02-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus (SLE); Immune-mediated Necrotizing Myopathy (IMNM); Neuromyelitis Optica Spectrum Disorders (NMOSD); Multiple Sclerosis (MS); Myasthenia Gravis; Systemic Sclerosis (SSc)
Keywords: CD20/BCMA-directed CAR-T cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Neuromyelitis Optica; Multiple Sclerosis; Myasthenia Gravis; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR168 (Experimental): Autologous C-CAR168 administered by intravenous (IV) infusion
  Interventions: Biological: CD20/BCMA-directed CAR-T cells

INTERVENTIONS:
Biological: CD20/BCMA-directed CAR-T cells — Autologous 2nd generation CD20/BCMA-directed CAR-T cells, single infusion intravenously
  Other Names: C-CAR168

SUMMARY:
This is an investigator-initiated, multicenter, open-label study of C-CAR168, an autologous bi-specific CAR-T therapy targeting CD20 and BCMA, for the treatment of adult patients with autoimmune diseases refractory to standard therapy

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old at the time of signing the Informed Consent Form (ICF).
* Diagnosed as SLE/Immune-Mediated Necrotizing Myopathy (IMNM)/Neuromyelitis Optica Spectrum Disorders (NMOSD)/Multiple Sclerosis (MS)/Myasthenia Gravis (MG)/Systemic Sclerosis (SSc) according to recognized diagnostic criteria for at least 6 months.
* Remains disease active or relapses after treatment with standard of care therapy for at least 8 weeks with the dose stable for more than 2 weeks; patients should have been treated with at least two immunosuppressants (including immunosuppressants, biologics, and disease-modifying drug (DMD) ).
* Adequate bone marrow, coagulation, cardiopulmonary, liver and renal function.

Exclusion Criteria:

* Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV), Treponema Pallidum (TP) positive, Cytomegalovirus (CMV) DNA positive, Epstein-Barr Virus (EBV) DNA positive.
* Uncontrolled active infection.
* Live vaccine injection within 4 weeks prior to signing the ICF.
* Major organ transplantation history or bone marrow/hematopoietic stem cell transplantation history.
* Severe cardiovascular diseases within the past 6 months prior to screening.
* ≥ Grade 2 bleeding within the past 30 days prior to screening, or requiring long-term anticoagulants treatment.
* Inadequate washing time for previous treatment.
* Previously treated with CAR-T cell products or genetically modified T cell therapies.
* Pregnant or lactating women.
* Severe central nervous system diseases or pathological changes.
* Malignancy history within 5 years prior to signing the ICF.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2040-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | Throughout the first 24 months follow up period completion (3 years)，DLTs will be observed/collected throughout the 28 days post C-CAR168 infusion
  Incidence of any adverse events (AEs), including dose limiting toxicities (DLTs)
The subsequent recommended dose of C-CAR168 in patients with autoimmune diseases refractory to standard therapy | Throughout the first 24 months follow up period completion (3 years)
  Based on the assessment of dose-limiting toxicities (DLTs) rates and overall safety profile

SECONDARY OUTCOMES:
The proportion of subjects who achieved remission at 6 months (6M) | Throughout the first 6 months follow up period completion (1.5 years)
The proportion of subjects who achieved remission during the main study period | Throughout the first 24 months follow up period completion (3 years)
The proportion of subjects who experienced relapse during the main study period | Throughout the first 24 months follow up period completion (3 years)
Time to response (TTR) | Throughout the first 24 months follow up period completion (3 years)
  The time from the date of C-CAR168 infusion to the first documented remission
Progression-free survival (PFS) | Throughout the first 24 months follow up period completion (3 years)
  The time from the date of C-CAR168 infusion to the date of first documented disease progression or death, whichever comes first
The proportion of subjects who achieved glucocorticoids/immunosuppressant free and subjects who achieved low-dose glucocorticoids application during the main study period | Throughout the first 24 months follow up period completion (3 years)
Maximal plasma concentration (Cmax) | Throughout the first 24 months follow up period completion (3 years)
  Maximal plasma concentration of C-CAR168 in peripheral blood
Time to reach the maximal plasma concentration (Tmax) | Throughout the first 24 months follow up period completion (3 years)
  Time to reach the maximal plasma concentration of C-CAR168 in peripheral blood
Duration in peripheral blood (Tlast) | Throughout the first 24 months follow up period completion (3 years)
  The duration of C-CAR168 in peripheral blood
Area under curve (AUC) | Throughout the first 24 months follow up period completion (3 years)
  Area under the curve of C-CAR168 in peripheral blood
The clearance of peripheral blood B cell | Throughout the first 24 months follow up period completion (3 years)
The decline of serum immunoglobulin | Throughout the first 24 months follow up period completion (3 years)
The elevation of peripheral blood complement | Throughout the first 24 months follow up period completion (3 years)
The decline of autoantibodies or other disease specific biomarkers | Throughout the first 24 months follow up period completion (3 years)

OTHER OUTCOMES:
Serum cytokines (including Interleukin (IL)-2, IL-4, IL-6, IL-10, Tumor Necrosis Factor (TNF)-α, Interferon (IFN)-γ) changes | Throughout the first 24 months follow up period completion (3 years)
  Detection of serum cytokines (including IL-2, IL-4, IL-6, IL-10, TNF-α, IFN-γ) changes over time by flow cytometry
Soluble BCMA changes in peripheral blood | Throughout the first 24 months follow up period completion (3 years)
  Detection of soluble BCMA changes in peripheral blood by Enzyme Linked ImmunoSorbent Assay (ELISA)
RNA changes in peripheral blood | Throughout the first 24 months follow up period completion (3 years)
  Detection of RNA changes in peripheral blood by RNA sequencing
Protective antibodies changes in peripheral blood | Throughout the first 24 months follow up period completion (3 years)
  Detection of protective antibodies changes in peripheral blood by ELISA
B cells changes in bone marrow, skin, muscle or kidney | Throughout the first 24 months follow up period completion (3 years)
  Detection of B cells concentration changes in bone marrow, skin, muscle or kidney by flow cytometry
Plasma cells or long-lived plasma cells changes in bone marrow, skin, muscle or kidney | Throughout the first 24 months follow up period completion (3 years)
  Detection of plasma cells or long-lived plasma cells concentration changes in bone marrow, skin, muscle or kidney by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Nan Shen, MD & PhD, Principal Investigator — Department of Rheumatology, RenJi Hospital, School of Medicine, Shanghai JiaoTong University
Locations (1):
- Department of Rheumatology, RenJi Hospital, School of Medicine, Shanghai JiaoTong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No